CLINICAL TRIAL: NCT01110460
Title: Cross-sectional and Prospective Observational Study Aimed to Assess the Prevalence of Uncontrolled and Partially Controlled Asthmatics in Italy and the Prevalence of Uncontrolled/Partially Controlled Patients Achieved Asthma Control After 12 Months
Brief Title: Prospective Study on Asthma Control
Acronym: PRISMA
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Medidata Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PRISMA
Record Dates: First submitted 2010-04-23; First posted 2010-04-26 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Accordingly, the new update of the Global Initiative for Asthma (GINA) guidelines 2006 is based on the control of the disease and attempts to quantify and graduate the level of control by using a classification of asthmatic subjects into controlled,partly controlled and uncontrolled groups.

Achieving and maintaining optimal asthma control is a major goal of asthma management. Although the results of clinical trials advocate that asthma control can be reached in most patients, there is evidence that many subjects with asthma have poorly controlled disease and that there is a significant gap between the treatment goals and the current level of asthma control achieved in the general population.

The aim of this study is to assess the prevalence of uncontrolled and partly controlled asthma in Italy using a patient-based tool such as Asthma Control Test.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Male or female patients with asthma diagnosis (at least 6 months)
* ability to understand and fill in questionaires

Exclusion Criteria:

* Patients included in a clinical trial within the last 12 weeks
* Patients with serious illnesses
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients
Sampling Method: Probability Sample
Enrollment: 2875 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Asthma control test score | 3 months

SECONDARY OUTCOMES:
EuroQoL test score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Terzano, Study Director — Policlinico Umberto I Roma

REFERENCES:
- [Derived] Terzano C, Cremonesi G, Girbino G, Ingrassia E, Marsico S, Nicolini G, Allegra L; PRISMA (PRospectIve Study on asthMA control) Study Group. 1-year prospective real life monitoring of asthma control and quality of life in Italy. Respir Res. 2012 Dec 6;13(1):112. doi: 10.1186/1465-9921-13-112. PMID 23216798